CLINICAL TRIAL: NCT04812431
Title: A Single Center, Open Label, Single Group, Phase 1/2a Clinical Study to Evaluate the Safety and Exploratory Efficacy of Transplantation Therapy Using PSA-NCAM(+) NPC Derived From hESC Line in AIS-A Level of Sub-acute SCI(From 7 to 60 Days)
Brief Title: Safety and Exploratory Efficacy of Transplantation Therapy Using PSA-NCAM(+) NPC in AIS-A Level of Sub-acute SCI
Acronym: SB-SCI-001
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: S.Biomedics Co., Ltd. (Industry)
Collaborators: Linical Co., Ltd. (Industry); Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HI20C0168000020
Record Dates: First submitted 2021-02-24; First posted 2021-03-23 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injury, Acute; Spinal Cord Injury at C4 Level With Complete Lesion; Spinal Cord Injury at C5-C7 Level With Complete Lesion
Keywords: Spinal cord injury; AIS-A
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: All subjects with damage to C4-C7 cords diagnosed as AIS-A are administered with PSA-NCAM(+) NPC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PSA-NCAM(+) NPC (Experimental): Cells are administered through intrathecal injection. Injection is administered to a total of five areas.
  Interventions: Biological: Neural precursor cells derived from human embryonic stem cell line

INTERVENTIONS:
Biological: Neural precursor cells derived from human embryonic stem cell line — When the Dose Limiting Toxicity (DLT) is not presented in the first three subjects administered with PSA-NCAM(+) NPC, two additional patients are added to the clinical study.

SUMMARY:
This study intends to evaluate the safety and exploratory efficacy of transplantation therapy using neural precursor cells (PSA-NCAM(+) NPC) derived from the human embryonic stem cell line for the treatment of paralysis and other related symptoms from sub-acute spinal cord injury.

DETAILED DESCRIPTION:
Subjects with damage to C4-C7 cords diagnosed as AIS-A are administered with PSA-NCAM(+) NPC.

For evaluation of safety and exploratory efficacy, 2 to 6 subjects will be enrolled depending on the presentation of dose-limiting toxicity.

When the Dose Limiting Toxicity (DLT) is not presented in the first three subjects administered with PSA-NCAM(+) NPC, two additional patients are added to the clinical study. When the DLT is presented in two or more of the first three patients, the clinical study is discontinued; when the DLT is presented in one of the three patients, three additional new patients are added. In case of presentation of the DLT in at least one of the three additional patients, the study is discontinued; the clinical study is continued only when the DLT is not presented in all three patients.

Screening visit (Visit 1), surgery and recovery visit (Visit 2 to Visit 6), follow-up visit (Visit 7 to Visit 8 + phone screening I, II, III), additional visit (Visit 9 to Visit 10), and close-out visit (Visit 11) are conducted. A clinical study period of at least 68 weeks is secured after Visit 6 (at least 5 visits and 3 phone screenings).

All subjects are to be conducted of follow-up study of a period of 1 year and 5 months at Weeks 1, 2, 4, 8, 12, 24, 48, and 72 after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Upon written consent of the patient or the legally acceptable representative of the patient
2. Male and female patients 18 to 65 years of age
3. Female patients who showed negative results on the pregnancy test, use an acceptable contraceptive or have no possibility of pregnancy (at least 2 years have elapsed after menopause or have undergone hysterectomy, ovariectomy, or sterilization operation), or male patients who have received vasectomy or are willing to use contraceptives for up to 90 days after administration of the investigational product using a dual contraceptive method*

   *Dual contraceptive method: Method of using multiple contraceptives, such as using a cervical cap or contraceptive diaphragm in addition to a condom for males
4. Patients who are capable of being administered with the investigational product on Day 7 to 60 after spinal cord injury
5. Patients who have been confirmed to have spinal cord injury classified as AIS-A on ISNCSCI, SCIM and/or MRI by the investigator, physiatrist, or other spinal cord injury specialist
6. Patients whose ASIA Impairment Scale (AIS) satisfies AIS-A criteria (spinal segment within C4-C7, complete injury)

Exclusion Criteria:

1. Patients with spinal cord injury caused by penetrating trauma such as gunshot or stab wounds
2. Patients with complete transection on the spinal cord
3. Patients with spinal cord injury that require more than the mono-segment treatment
4. Patients with other complications, including neurological defects related to peripheral nerve injury (neuromuscular injury or central spinal cord syndrome), or etiological causes of paraplegia or sensorimotor defects related to an additional underlying condition
5. Patients with multiple lesions or lesions longer than 2 cm in length found on MRI examination
6. Patients administered with cells excluding blood transfusion before participating in the clinical study
7. Patients with the following intercurrent diseases or conditions:

   1. Coagulopathy with INR> 1.4 at the time of administration of the investigational product (Day 0)
   2. Active infection
   3. Active hypotension requiring vasoconstrictor treatment (less than 60 mmHg of diastolic blood pressure)
   4. Rupture of the skin on the area of surgery
   5. Medical history of malignant tumor
   6. Primary or secondary immunodeficiency
   7. Clinically significant abnormal values discovered as a result of laboratory tests

      * Creatinine > 1.5 mg/dL
      * When the level found in the liver-function examination is more than twice the upper limit of the normal level
      * Hematocrit/hemoglobin <30%/10 g/dL
      * Total WBC < 1000/μL
      * Uncontrolled hypertension (systole> 180 mmHg or diastole> 100 mmHg)
      * Uncontrolled diabetes (HbA1c> 8%)
      * Evidence of GI bleeding on the stool guaiac test
      * Positive on tuberculosis test (However, a chest X-ray may be performed if found positive on the TB test, and the patient may be enrolled upon no findings that suggest active tuberculosis on the chest X-ray.)
      * Hepatitis B or C
      * Human Immunodeficiency Virus (HIV)
   8. Substance abuse or alcoholism
   9. Unstable or untreated psychiatric disorder
8. Patients with known hypersensitivity to basiliximab, tacrolimus, mycophenolate mofetil, methylprednisolone, or prednisone
9. Patients incapable of receiving physical therapy or combination therapy
10. Patients incapable of going under general anesthesia due to other reasons
11. Patients judged unsuitable for participation in this clinical study by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Changes of occurred adverse events during the clinical study | Visit 3(Day 0), Visit 4(1 week), Visit 5(2 weeks), Visit 6(4 weeks), Visit 7(8 weeks), Visit 8(12 weeks), Visit 9(24 weeks), Visit 10(48 weeks), Visit 11(72 weeks), Telephone visit 1(13 weeks), Telephone visit 2(14 weeks), Telephone visit 3(16 weeks)
  Assessment of the presentation rate of adverse events occurred from IP administration until the end of the clinical study (Visit 11).
Rate of abnormal signs as assessed through physical examination | Visit 1(Screening), Visit 11(72 weeks)
  Assessment of the normal/abnormal changes at the baseline (Visit 1) and changes at the end of the clinical study (Visit 11) as assessed through physical examination (appearance, skin, head/neck, chest/lung, heart, abdomen, genitourinary system, extremities, musculoskeletal system, nervous system, and lymph nodes).
Measured changes of Systolic blood pressure (mm Hg) | Visit 1(Screening), Visit 2(-2 Day), Visit 3(Day 0), Visit 4(1 week), Visit 5(2 weeks), Visit 6(4 weeks), Visit 7(8 weeks), Visit 8(12 weeks), Visit 9(24 weeks), Visit 10(48 weeks), Visit 11(72 weeks)
  Comparative assessment of measured value using systolic blood pressure (mm Hg) from the baseline (Visit 1) to the end of the clinical study (Visit 11).
Measured changes of Body temperature (degrees Celsius) | Visit 1(Screening), Visit 2(-2 Day), Visit 3(Day 0), Visit 4(1 week), Visit 5(2 weeks), Visit 6(4 weeks), Visit 7(8 weeks), Visit 8(12 weeks), Visit 9(24 weeks), Visit 10(48 weeks), Visit 11(72 weeks)
  Comparative assessment of measured value using body temperature (degrees Celsius) from the baseline (Visit 1) to the end of the clinical study (Visit 11).
Measured changes of Heart rate (beats per minute) | Visit 1(Screening), Visit 2(-2 Day), Visit 3(Day 0), Visit 4(1 week), Visit 5(2 weeks), Visit 6(4 weeks), Visit 7(8 weeks), Visit 8(12 weeks), Visit 9(24 weeks), Visit 10(48 weeks), Visit 11(72 weeks)
  Comparative assessment of measured value using heart rate (beats per minute) from the baseline (Visit 1) to the end of the clinical study (Visit 11).
Measured changes of Respiratory rate (breaths per minute) | Visit 1(Screening), Visit 2(-2 Day), Visit 3(Day 0), Visit 4(1 week), Visit 5(2 weeks), Visit 6(4 weeks), Visit 7(8 weeks), Visit 8(12 weeks), Visit 9(24 weeks), Visit 10(48 weeks), Visit 11(72 weeks)
  Comparative assessment of measured value using respiratory rate (breaths per minute) from the baseline (Visit 1) to the end of the clinical study (Visit 11).
Rate of abnormal hematology values | Visit 1(Screening), Visit 2(-2 Day), Visit 3(Day 0), Visit 4(1 week), Visit 5(2 weeks), Visit 6(4 weeks), Visit 7(8 weeks), Visit 8(12 weeks), Visit 9(24 weeks), Visit 10(48 weeks), Visit 11(72 weeks)
  Assessment of the normal/abnormal changes at the baseline (Visit 1) and changes at the end of the clinical study (Visit 11) as measured value using hematology values(WBC, WBC differential, RBC, Hemoglobin, Hematocrit, and Platelet).
Rate of abnormal chemistry values | Visit 1(Screening), Visit 2(-2 Day), Visit 3(Day 0), Visit 4(1 week), Visit 5(2 weeks), Visit 6(4 weeks), Visit 7(8 weeks), Visit 8(12 weeks), Visit 9(24 weeks), Visit 10(48 weeks), Visit 11(72 weeks)
  Assessment of the normal/abnormal changes at the baseline (Visit 1) and changes at the end of the clinical study (Visit 11) as measured value using chemistry values(Sodium, Potassium, Calcium, Chloride, Inorganic Phosphate, SGOT(AST), SGPT(ALT), Alkaline Phosphatase, GGT, Creatinine, BUN, Total Bilirubin, Total Protein, Albumin, and Glucose).
Rate of abnormal urinalysis values | Visit 1(Screening), Visit 2(-2 Day), Visit 3(Day 0), Visit 4(1 week), Visit 5(2 weeks), Visit 6(4 weeks), Visit 7(8 weeks), Visit 8(12 weeks), Visit 9(24 weeks), Visit 10(48 weeks), Visit 11(72 weeks)
  Assessment of the normal/abnormal changes at the baseline (Visit 1) and changes at the end of the clinical study (Visit 11) as measured value using urinalysis values(Protein, Glucose, Ketones, and Occult Blood).
Measured changes of diastolic blood pressure (mm Hg) | Visit 1(Screening), Visit 2(-2 Day), Visit 3(Day 0), Visit 4(1 week), Visit 5(2 weeks), Visit 6(4 weeks), Visit 7(8 weeks), Visit 8(12 weeks), Visit 9(24 weeks), Visit 10(48 weeks), Visit 11(72 weeks)
  Comparative assessment of measured value using diastolic blood pressure (mm Hg) from the baseline (Visit 1) to the end of the clinical study (Visit 11).

SECONDARY OUTCOMES:
Assessment of Graft survival at the transplant site as observed in MRI examination | Visit 1(Screening), Visit 11(72 weeks)
  Number of participants with measured value(spinal cord changes, spinal cord atrophy far from the lesion, edema, cystic degeneration, spinal sinus, and diameter change) using MRI examination.
Number of participants with Transplant rejection against transplanted cells | Visit 1(Screening), Visit 6(4 weeks)
  Comparative Assessment of PSA-NCAM(+) NPC-specific antibody that may result in transplant rejection in the HLA antigen/antibody reaction test.
Changes in the ASIA Damage Scale | Visit 1(Screening), Visit 8(12 weeks), Visit 11(72 weeks)
  Number of participants with changes in ISNCSCI ASIA at Week 12 (Visit 8) and Week 72 (Visit 11) of administration compared to the baseline (Visit 1).
International standards for neurological classification of spinal cord injury (ISNCSCI) motor index score | Visit 1(Screening), Visit 6(4 weeks), Visit 8(12 weeks), Visit 9(24 weeks), Visit 10(48 weeks), Visit 11(72 weeks)
  Number of participants with motor level recovered* at Week 4 (Visit 6), Week 12 (Visit 8), Week 24 (Visit 9), Week 48 (Visit 10), and Week 72 (Visit 11) of drug administration compared to the baseline (Visit 1).
  * Recovery: Subjects with recovery of at least 2 stages in the upper limb motor score
Measured changes of International standards for neurological classification of spinal cord injury (ISNCSCI) sensory index score | Visit 1(Screening), Visit 8(12 weeks), Visit 11(72 weeks)
  Rate of changes in the total ISNCSCI ASIA sensory index score at Week 12 (Visit 8) and Week 72 (Visit 11) of administration compared to the baseline (Visit 1).
Pain assessment | Visit 1(Screening), Visit 8(12 weeks), Visit 11(72 weeks)
  Rate of measured changes in the pain scores at Week 12 (Visit 8) and Week 72 (Visit 11) compared to the baseline (Visit 1).
Spinal Cord Independence Measure (SCIM) score | Visit 1(Screening), Visit 8(12 weeks), Visit 11(72 weeks)
  Rate of change in the SCIM score at Week 12 (Visit 8) and Week 72 (Visit 11) compared to the baseline (Visit 1).
Measured changes of International standards for neurological classification of spinal cord injury (ISNCSCI) motor index score | Visit 1(Screening), Visit 8(12 weeks), Visit 11(72 weeks)
  Rate of changes in the total ISNCSCI ASIA motor score at Week 12 (Visit 8) and Week 72 (Visit 11) of administration compared to the baseline (Visit 1).

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ah Shin, MD, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (2):
- South Korea (2):
  - Ajou University Hospital, Suwon, Gyeonggido
  - Yonsei University Health System, Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No